CLINICAL TRIAL: NCT02026804
Title: Prevalence ， Associated Factors and Influences of Prenatal Mental Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial Natural Science Foundation of China (Other)
Responsible Party: Sponsor
Other Study IDs: Y21000505
Record Dates: First submitted 2013-12-30; First posted 2014-01-03 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Mental Disorder During Pregnancy - Baby Not Yet Delivered

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, white cells, placenta tissue

GROUPS / COHORTS (1):
- Prenatal mental disorders

SUMMARY:
The purpose of this study is to find the incidence of mental disorders during different periods of pregnancy and its associated factors and consequences.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years of age
* 8 to 12 weeks of pregnancy
* There is no history of mental illness
* Had perinatal health care in a Women's & Children's Health Hospital

Exclusion Criteria:

* The obvious body disease
* Having anxiety, phobia, hypochondriasis, obsessive-compulsive disorder or depression before pregnancy
* Having severe complications during pregnancy
* Fetal malformation or abortion
* Can't understand the questionnaire
* Without informed consent
* More than 13 weeks of pregnancy
* Less than 18 years of age

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who had perinatal health care in a Women's & Children's Health Hospital of zhejiang province, China
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of mental disorders during different periods of pregnancy | from 8 weeks of pregnancy to delivery
  We would like to find the incidence of mental disorders in early (8-12 weeks),middle (18-22 weeks) and later(32 weeks to delivery) period of pregnancy

SECONDARY OUTCOMES:
pregnancy outcomes | from 8 weeks of pregnancy to 6 months after delivery
  We would like to explore which period of mental disorders had the most significant infuences on pregnancy outcomes including obstetrical complications(e.g.gestational diabetes mellitus(GDM),hypertensive disorder complicating pregnancy(HDCP)),outcome of fetus(e.g.preterm,low birth weight and fetal anomaly) and health of infant and puerpera.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhoushan Women's & Children's Health Hospital, Zhoushan, Zhejiang, China